CLINICAL TRIAL: NCT06114810
Title: Immunogenicity of Novel Oral Poliovirus Vaccine Type 2 (nOPV2), Bivalent Oral Poliovirus Vaccine (bOPV) and Inactivated Poliovirus Vaccine (IPV) Administered With Different Sequential or Combination Schedules
Brief Title: Immunogenicity of Novel Oral Poliovirus Vaccine Type 2 (nOPV2), bOPV and IPV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Government of Bangladesh (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PR-23036
Record Dates: First submitted 2023-10-12; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-09

CONDITIONS: Polio
Keywords: nOPV2 bOPV IPV immunogenicity
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Intervention Model Description: This is an open-label, controlled, inequality, 4 arm randomized clinical trial assessing immunogenicity of several poliovirus vaccines and doses
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A : 3 doses of nOPV2 and bOPV with IPV (Active Comparator): Participants in arm A will receive the following polio vaccines: nOPV2 +bOPV (2 drops = 0.1 ml) @ 6, 10, 14 weeks and IPV (0.5 mL) @ 14 weeks
  Interventions: Biological: polio vaccines: nOPV2, bOPV, IPV
- Arm B : 2 doses of nOPV2 and bOPV with IPV (Active Comparator): Participants in arm B will receive the following polio vaccines: nOPV2+bOPV , (2 drops = 0.1 ml) @ 6, 10 weeks and IPV (0.5 mL) @ 14 weeks
  Interventions: Biological: polio vaccines: nOPV2, bOPV, IPV
- Arm C: Single dose of bOPV, nOPV2, IPV (Active Comparator): Participants in arm C will receive the following polio vaccines: bOPV ( 2 drops) @ 6 week , nOPV2 (2 drops) at 10 weeks and IPV ( 0.5mL) @ 14 weeks
  Interventions: Biological: polio vaccines: nOPV2, bOPV, IPV
- Arm D: Single dose nOPV2, IPV (Active Comparator): Participants in arm D will receive the following polio vaccines: nOPV2 (2 drops = 0.1 ml) at 6 and 10 weeks and IPV ( 0.5mL) @ 14 weeks
  Interventions: Biological: polio vaccines: nOPV2, bOPV, IPV

INTERVENTIONS:
Biological: polio vaccines: nOPV2, bOPV, IPV — Co-administration of nOPV2 with bOPV along with IPV with different sequential or combination schedules.

SUMMARY:
The goal of this clinical trial is to explore two strategies to enhance nOPV2 immunogenicity in the field and overcome potential interference of bOPV:

1. Addition of IPV after one or several doses of nOPV2 and bOPV to close remaining immunity gaps;
2. Separation of bOPV and nOPV2 with an interval of 4 weeks.

Participants at 6 weeks of age will be enrolled and randomized to one of four arms receiving the different polio vaccines; nOPV2, bOPV and IPV, in different combination schedule. The target enrolment is 220 infants per arm for a total of 880. Blood will be collected from all participants to measure Poliovirus antibody titers to types 1, 2 and 3.

DETAILED DESCRIPTION:
The study will assess whether adding IPV at the end of a 3-dose series of co-administered nOPV2+bOPV achieves at least a 95% seroconversion to all serotypes and whether adding IPV following two doses of co-administered nOPV2+bOPV achieves at least a 90% seroconversion to all poliovirus types.

Study findings will inform vaccination strategies in areas with co-circulation of poliovirus types and provide information about immunogenicity of potential routine immunization schedule with nOPV2 and bOPV in countries with persistent transmission or emergences of cVDPV2.

This is an open-label, controlled, inequality, four arm randomized clinical trial, will be conducted in two study sites in Dhaka, Bangladesh. Participants will be enrolled at 6 weeks of age following inclusion and exclusion criteria's, randomly assigned to one of the four study arms and followed to 18 weeks of age. Three polio vaccines will be used in the study: bOPV, nOPV2 and IPV in different sequential or combination schedules.

Entry evaluations will be completed at 6 weeks of age. Blood collection and study vaccine administration are planned during the study entry evaluation. Post-entry evaluations and follow-up will be done at 10 weeks, 14 weeks and 18 weeks of age. Blood will be collected before any study or EPI vaccines are administered. Presence of poliovirus neutralizing antibodies to all three poliovirus types will be assessed using a microneutralization assay.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants 6 weeks of age
2. Parents that consent for participation in the full length of the study.
3. Parents that can understand and comply with planned study procedures.

Exclusion Criteria:

1. Parents and infants are unable to participate in the full length of the study
2. A diagnosis or suspicion of immunodeficiency disorder either in the infant or in an immediate family member.
3. A diagnosis or suspicion of bleeding disorder
4. Acute diarrhoea, infection, or illness at the time of enrolment
5. Acute vomiting and intolerance to liquids within 24 hours before the enrolment visit
6. Evidence of a chronic medical condition
7. Receipt of any polio vaccine (OPV or IPV) before enrolment
8. Known allergy/sensitivity or reaction to polio vaccine, or its contents.
9. Infants from multiple births.
10. Infants from premature births (<37 weeks of gestation).

Ages: 42 Days to 48 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 880 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Cumulative seroconversion to all serotypes at the end of a vaccination series including two or three doses of co-administered nOPV2 and bOPV plus one dose of IPV. | Serology: 6 &18 weeks
  Poliovirus antibody titers to types 1, 2 and 3 will be measured in sera extracted from blood collected at 6, 10, 14, and 18 weeks of age

SECONDARY OUTCOMES:
Seroconversion for type 2 after one dose of nOPV2 alone, co-administered with bOPV, or administered 4-weeks after bOPV; | Serology: 6 & 14 weeks for C, 6 & 10 weeks for D,
  Compare type 2 seroconversion after one dose of nOPV2 administered alone or 4 weeks after bOPV
Cumulative seroconversion for type 2 after two doses of nOPV2 administered alone or co-administered with bOPV; | Serology: 6 & 14 weeks for C, 6 & 10 weeks for A
  Compare seroconversion to all three serotypes after one dose of nOPV2 administered 4 weeks after bOPV or concomitantly with bOPV
Cumulative seroconversion to all serotypes after 1 dose each of bOPV, nOPV2 and IPV administered sequentially one month apart. | Serology: 6 & 18 weeks
  Determine seroconversion to all serotypes reached with one dose of nOPV2, bOPV and IPV each administered sequentially at 4-week intervals (6, 10 and 14 weeks).
Antibody titers for all 3 serotypes reached at the end of each vaccination schedule | Serology: 6 & 18 weeks
  Determine seroconversion to all serotypes

CONTACTS AND LOCATIONS:
Overall Officials: Dr. K Zaman, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
Study data will be jointly owned by icddr,b and CDC. After completion of study activities, summary tables of study results will be available on www.clinicaltrials.gov. After study registration, clinicaltrials.gov provides unrestricted public access on study details including summary tables.
  Study investigators will have access to all participants' data without identifiers, including laboratory data. Co-investigators and technical advisors will have access to relevant data as defined in protocol
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After study registration, clinicaltrials.gov. provides unrestricted public access on study details including summary tables.
  After completion of study activities, summary tables of study results will be available on www.clinicaltrials.gov.
  Study investigators will have access to all participants' data without identifiers, including laboratory data.
Access Criteria: Log in www.clinicaltrials.gov